CLINICAL TRIAL: NCT04664634
Title: A Digital Therapeutic Platform for Swallowing and Drooling Problems in Parkinson's
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Shuai (Steve) Xu, Principal Investigator, Northwestern University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: STU00221904
Record Dates: First submitted 2020-12-06; First posted 2020-12-11 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Dysphagia; Parkinson Disease
MeSH Terms: conditions — Deglutition Disorders; Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single Arm (Experimental): The Aria sensor is a wearable patch that continuously monitors physiological signals and provides vibratory haptic cues to increase swallow frequency. The intervention consists of using the sensor over a 3-week period, with active haptic cueing during Week 2 only.
  Interventions: Device: Aria Sensor

INTERVENTIONS:
Device: Aria Sensor — The Aria sensor is a wearable patch that continuously monitors physiological signals and provides vibratory haptic cues to increase swallow frequency. The intervention consists of using the sensor over a 3-week period, with active haptic cueing during Week 2 only.

SUMMARY:
The purpose of this study is the development and early-stage validation of a wearable sensor for dysphagia in patients with PD.

DETAILED DESCRIPTION:
The project goal is the development and early stage validation of a wearable sensor for dysphagia in patients with PD. The first phase of the program involves engineering goals relating to increasing the battery life of this sensor to 48 hours between charges and reducing the overall form factor size. The second phase of the program is to conduct focus groups with PD patients to assess sensor usability, set up burden, and design feedback. The third phase of the study will assess the feasibility of the sensor to detect and cue swallowing in a small cohort of PD patients.

ELIGIBILITY:
Inclusion criteria. Age ≥22. English speaking. Diagnosis of idiopathic Parkinson's disease of any Hoehn and Yahr stage (I-V), determined by a neurologist.

Mild to moderate sialorrhea defined as a score of ≥ 11* on the Radboud Oral Motor Inventory for Parkinson's Disease (ROMP)-Saliva (C) subscale Subjects must be in the "on" phase of their medication during all study assessments. The "on" phase is defined as the period when the participant's medication is at peak effectiveness, minimizing motor fluctuations and enabling optimal motor function.

Study Exclusion Criteria. History of aspiration pneumonia within the past 12 months. Unable to swallow saliva without a maneuver. Actively receiving treatment for swallowing disorders or sialorrhea. Current alcohol/drug abuse. Diagnosed with neurological disorders other than PD. End stage dementia. History of head and neck cancer or surgery. Unable to demonstrate competency with the user-friendly sensor platform technology.

Known allergy to contrast material used during MBSS. Known allergy to sensor adhesive. Indwelling tracheostomy tube. Nasogastric (NG) feeding tube. Currently pregnant.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Percent agreement with Gold Standard | 1 year
  Percent agreement between experimental sensor Gold standard (GS) respiratory inductance plethysmography (RIP) with Inductotrace System®, Ambulatory Monitoring)
Change in mean swallow frequency during haptic cueing week | Week 1 to Week 2
  This outcome measures the change in the average number of swallows per hour during the intervention week (Week 2, with haptic cueing) compared to baseline (Week 1, no cueing). Swallows will be manually labeled from sensor audio recordings by at least three independent annotators.

SECONDARY OUTCOMES:
Change in algorithm-detected swallow frequency during haptic cueing week | Week 1 to Week 2
  This outcome measures the change in the mean swallow frequency as automatically detected by the Aria sensor's AI algorithm, comparing Week 2 (intervention) to Week 1 (baseline). Performance will be benchmarked against manually annotated swallows.
Change in Sialorrhea Clinical Scale for Parkinson's Disease (SCS-PD) score | Baseline to Week 3
  Assesses the effect of the intervention on drooling symptoms using the Sialorrhea Clinical Scale for PD. Participants complete this validated questionnaire at baseline, during, and after the intervention.
Change in ROMP-Swallowing Subscale score | Baseline to Week 3
  Assesses changes in self-reported swallowing function using the Swallowing Subscale of the Radboud Oral Motor Inventory for Parkinson's Disease (ROMP). The ROMP is a validated, PD-specific measure.
Change in participant adherence to haptic cueing | Week 2
  Evaluates adherence to the intervention by quantifying the percentage of haptic cues that are followed by a swallow within 5 seconds during Week 2. Cue-swallow pairings are based on algorithmic and manual labeling.

OTHER OUTCOMES:
Change in Modified Barium Swallow Impairment Profile (MBSImP) | Baseline to Week 3
  Subsample of participants will undergo video fluoroscopy to evaluate swallowing function. The MBSImP scores will assess changes in swallow physiology pre- and post-intervention.
Change in Penetration-Aspiration Scale Score | Baseline to Week 3
  Assesses airway protection during swallowing via penetration-aspiration scale scores from videofluoroscopic studies in a subsample of participants.

CONTACTS AND LOCATIONS:
Locations (1):
- Northwestern University, Evanston, Illinois, United States